CLINICAL TRIAL: NCT04284059
Title: Adjuvant Effects of Vitamin A and Vitamin D Supplementation on Treatment of Children With ADHD:A Randomized, Double Blind, Placebo-controlled, Multicentric Trial.
Brief Title: Adjuvant Effects of Vitamin A and Vitamin D Supplementation on Treatment of Children With ADHD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chen Li (Other)
Responsible Party: Sponsor-Investigator, Chen Li, Associate Professor，Director, Children's Hospital of Chongqing Medical University
Organization: Children's Hospital of Chongqing Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CHENLI
Record Dates: First submitted 2020-02-20; First posted 2020-02-25 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: ADHD
Keywords: Vitamin A; Vitamin D; Methylphenidate; ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Vitamin D

STUDY DESIGN:
Intervention Model Description: The patients showed deficiency or insufficiency in vitamin A (≤1.05 umol/ L) and vitamin D (≤50 nmol/L) are randomly assigned in double-blind fashion in a 1:1:1 ratio to the vitamin AD supplementation group, vitamin D supplementation group or the placebo group. Vitamin AD supplementation group will be administrated vitamin AD capsules (3 capsules/time, once a day for 8 weeks), which contain vitamin A (2000 IU/capsule) and vitamin D (700 IU/capsule). Vitamin D supplementation group will be administrated vitamin D capsules (400 IU/capsule, 6 capsules/time, once a day for 2 weeks, then change to 5 capsules/time, once a day for 6 weeks). The placebo capsules given to the placebo group (3 capsules/time, once a day for 8 weeks), consists of oily liquids which do not contain vitamin A and vitamin D, and were produced in strict accordance with China's drug management and packaging requirements for placebo by Shandong DYNE Marine Biopharmaceutical Co., Ltd in China.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The participants and care providers don't know which group they are enrolled in. And the investigators just play a roll in recruiting the patients, inform the patients about the study, and then randomly assign the patients in a 1:1:1 ratio to the A group, B group or C group. The drugs are dispensed by staff who was not involved in the process of evaluation, diagnosis and treatment. The staff will take notes about the patients' basic information and medication records. After the study, the staff will give the unblinded results to to investigators and outcomes assessor. The investigators will provide the compensatory therapy for the patients. The outcomes assessor will do the statistic analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- vitamin AD group (Active Comparator): The patients aged 6-12 with a diagnose of ADHD of this group is deficient or insufficient in vitamin A and vitamin D. They will receive vitamin A 6000 IU/day and vitamin D 2100 IU/day supplementation in addition to methylphenidate for 8 weeks.
  Interventions: Dietary Supplement: vitamin AD
- vitamin D group (Experimental): The patients aged 6-12 with a diagnose of ADHD of this group is deficient or insufficient in vitamin A and vitamin D. They will receive vitamin D 2100 IU/day supplementation in addition to methylphenidate for 8 weeks. After the study, vitamin D group will be administrated with vitamin A on the basis of serum retinol concentration after the study.
  Interventions: Dietary Supplement: vitamin D
- placebo group (Placebo Comparator): The patients aged 6-12 with a diagnose of ADHD of this group is deficient or insufficient in vitamin A and vitamin D. They will receive placebo once a day in addition to methylphenidate for 8 weeks. After the study, the placebo group will be prescribed with vitamin A and vitamin D supplementation on the grounds of retinol and 25 (OH)D concentration.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Placebos — Placebo, vitamin AD and vitamin D are identical in the appearance to guarantee blind. The patients need to administrate 3 capsules once a day for 8 weeks.
  Arms: placebo group
Dietary Supplement: vitamin AD — A vitamin AD capsule contains vitamin A 2000 IU and vitamin D 700 IU. The patients need to administrate 3 capsules once a day for 8 weeks.
  Arms: vitamin AD group
Dietary Supplement: vitamin D — A vitamin D capsule contains vitamin D 400 IU. The patients need to asministrate 6 capsules/time, once a day for 2 weeks, then change to 5 capsules/time, once a day for 6 weeks.
  Arms: vitamin D group

SUMMARY:
Around 7.2% of children around the world are suffering from ADHD. On account of current medical treatment, a high remission rate can be reached for ADHD. Nevertheless, patients have to face a number of side effects associated with the treatment. It was informed that patients of ADHD have a tendency to vitamin A and vitamin D deficiency. The aim of the study is to determine the effect of vitamin A and vitamin D supplementation as adjunctive therapy to methylphenidate on symptoms of ADHD. 504 subjects aged 6-12 years with a diagnosis of ADHD based on DSM-5 criteria are randomly assigned into three groups to receive vitamin A 6000 IU/day and vitamin D 2100 IU/day, or vitamin D 2100 IU/day or placebo adding to methylphenidate for 8 weeks. Symptoms severity is assessed by Vanderbilt Assessment Scales and Questionnaire - Children with Difficulties at weeks 0, 4, and 8. Serum levels of retinol and 25(OH)D are measured at baseline and after 8 weeks. All the other sociodemographic data are assessed. The study can give more references on the application of vitamin A and vitamin D in addition to methylphenidate to ADHD. Future research is needed to clarify mechanism of vitamin A and vitamin D on ADHD.

DETAILED DESCRIPTION:
1. Procedures The patients showed deficiency or insufficiency in vitamin A (≤1.05 umol/ L) and vitamin D (≤50 nmol/L) are stratified by gender and randomly assigned in double-blind fashion in a 1:1:1 ratio to the vitamin AD supplementation group, vitamin D supplementation group or the placebo group. The participants will be given the related interventions. Placebo constituents by oily liquids without vitamin A and vitamin D. Placebo, vitamin AD and vitamin D are identical in the appearance to guarantee blind. These patients will be followed up at weeks 4 and 8 to evaluate the changes of ADHD symptoms after adding the adjunctive therapy to methylphenidate. And serum concentration of retinol and 25(OH)D are measured at weeks 8. Accordingly, the placebo group and vitamin D group will be prescribed with vitamin A and vitamin D supplementation on the grounds of retinol and 25 (OH)D concentration after the study.
2. Demographic questionnaire and clinical data The demographic questionnaire is completed by the child's primary caregiver, detailing child's name, gender, date of birth, height, weight, blood pressure, heart rate ; supplementation of vitamin A/D products or vitamin A/D-containing products. Clinical data will be ascertained from the medical records, including information about DSM-5 diagnosis, disease classification, current treatment, and comorbid conditions.
3. Sample size This study is a randomized double-blind controlled trial. Intervention groups are vitamin AD group and vitamin D group, control group is placebo group. The primary outcome index is changes in ADHD symptoms evaluated by Vanderbilt Assessment Scales and Questionnaire - Children with Difficulties (QCD) in the last 4 weeks or 8 weeks. The second outcome is the serum concentration of vitamin A and vitamin D. Conner's Parent Rating Scale (CPRS) was considered as the main outcome in the previous literature, the mean ± SD of ADHD index was 55.84 ± 10.2, 56.79 ± 9.6 for vitamin D + methylphenidate(n = 25), placebo + methylphenidate (n = 29) respectively. The investigators cautiously presume that the mean ± SD for vitamin AD + methylphenidate is 54 ± 9.88. Considering 0.05 of the alpha and 0.80 of power, a sample of 453 subjects divided among 3 groups are calculated by PASS 2020. And 504 subjects are enrolled in the study based on the dropout rate of 10%.
4. Statistical analysis All the data are analyzed using SPSS 19.0. The normality of variables are assessed by Kolmogorov Smirnov test. Comparison of parametric and nonparametric variables between groups are examined by F test and Kruskal-Wallis test, respectively. Paired t-test and Wilcoxon signed-rank test are used to investigate within-group differences. Confounding factors are adjusted by the analysis of covariance.
5. Bias control the investigators will describe both responders and non-responders on demographic questionnaire and clinical data in detail to assess the selection bias. And in order to decrease the dropout rate, the investigators will contact with the patient's parents about compliance to therapy by Wechat, E-mail, sometimes telephone contact is necessary.
6. Ethical matters and data protection The patients participated in the study will sign the informed consent (obtained from the guardian). And this study was approved by the local ethics committee . Patient's name will be abbreviated and the research data will be assigned a code then to provide to the researcher. The authorization from parents on the patient's health information remains valid until the study is completed. After that, researchers will delete private information from the study record.

ELIGIBILITY:
Inclusion Criteria:

* Diagnose of ADHD according to DSM-5
* Aged 6-12 years
* Intelligence quotient (IQ) ≥70
* Receiving methylphenidate (trade name Concerta) 18-54 mg/day once a day (began with 18 mg/day for a week and titrated gradually to the optimum dose not more than 54 mg/day).

Exclusion Criteria:

* Inconsistent or changing dose of methylphenidate during the participation period
* Use of anticonvulsant drugs or hydrocortisone
* Suffering from other neurological disorders and mental diseases now or in the past, such as convulsions, anxiety and depression
* Suffer from metabolic disorders such as cholestasis, liver dysfunction, pancreatic insufficiency, measles, diarrhea, respiratory illness, severe inflammation or malnutrition, etc.
* Use of vitamins and vitamin-containing products
* IQ≤70
* The serum concentration of vitamin A >1.05 umol/L and/ or vitamin D >50 nmol/L

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 504 (Estimated)
Dates: Start 2021-02-25 (Actual); Primary Completion 2022-05-30 (Estimated); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
The changes in ADHD clinical symptoms-Predominantly Inattentive subtype estimated by Chinese version of Vanderbilt parent assessment scale | at baseline
  The Vanderbilt parent assessment scale is designed to measure the severity of ADHD symptoms for children aged 6 to 12. It has 2 components: symptom assessment and impairment in performance. The symptom assessment screens for symptoms relevant to inattentive (items 1-9) and hyperactive (items 10-18) ADHD. The items 49-56 are performance measures. The symptom measures in the scale, scored 0 to 3. A positive response in symptom assessment part is a 2 or 3 (often, very often). The performance measures in the scale, scored 1 to 5, with 4 and 5 being somewhat of a problem/problematic.
  The scoring standard for Predominantly Inattentive subtype: Must score a 2 or 3 on 6 out of 9 items on questions 1-9 AND Score a 4 or 5 on any of the Performance questions 49-56. The higher scores mean a worse outcome.
The changes in ADHD clinical symptoms-Predominantly Inattentive subtype estimated by Chinese version of Vanderbilt teacher assessment scale | at baseline
  The Vanderbilt teacher assessment scale is designed to measure the severity of ADHD symptoms for children aged 6 to 12. It has 2 components: symptom assessment and impairment in performance. The symptom assessment screens for symptoms relevant to inattentive (items 1-9) and hyperactive (items 10-18) ADHD. The items 36-43 are performance measures. The symptom measures in the scale, scored 0 to 3. A positive response in symptom assessment part is a 2 or 3 (often, very often). The performance measures in the scale, scored 1 to 5, with 4 and 5 being somewhat of a problem/problematic.
  The scoring standard for Predominantly Inattentive subtype: Must score a 2 or 3 on 6 out of 9 items on questions 1-9 AND Score a 4 or 5 on any of the Performance questions 36-43. The higher scores mean a worse outcome.
The changes in ADHD clinical symptoms-Predominantly Hyperactive/Impulsive subtype estimated by Chinese version of Vanderbilt parent assessment scale | at baseline
  The Vanderbilt parent assessment scale is designed to measure the severity of ADHD symptoms for children aged 6 to 12. It has 2 components: symptom assessment and impairment in performance. The symptom assessment screens for symptoms relevant to inattentive (items 1-9) and hyperactive (items 10-18) ADHD. The items 49-56 are performance measures. The symptom measures in the scale, scored 0 to 3. A positive response in symptom assessment part is a 2 or 3 (often, very often). The performance measures in the scale, scored 1 to 5, with 4 and 5 being somewhat of a problem/problematic.
  The scoring standard for Predominantly Hyperactive/Impulsive subtype: Must score a 2 or 3 on 6 out of 9 items on questions 10-18 AND Score a 4 or 5 on any of the Performance questions 49-56. The higher scores mean a worse outcome.
The changes in ADHD clinical symptoms-Predominantly Hyperactive/Impulsive subtype estimated by Chinese version of Vanderbilt teacher assessment scale | at baseline
  The Vanderbilt teacher assessment scale is designed to measure the severity of ADHD symptoms for children aged 6 to 12. It has 2 components: symptom assessment and impairment in performance. The symptom assessment screens for symptoms relevant to inattentive (items 1-9) and hyperactive (items 10-18) ADHD. The items 36-43 are performance measures. The symptom measures in the scale, scored 0 to 3. A positive response in symptom assessment part is a 2 or 3 (often, very often). The performance measures in the scale, scored 1 to 5, with 4 and 5 being somewhat of a problem/problematic.
  The scoring standard for Predominantly Hyperactive/Impulsive subtype: Must score a 2 or 3 on 6 out of 9 items on questions 10-18 AND Score a 4 or 5 on any of the Performance questions 36-43. The higher scores mean a worse outcome.
The changes in ADHD clinical symptoms-ADHD Combined Inattention/Hyperactivity estimated by Chinese version of Vanderbilt parent assessment scale | at baseline
  The Vanderbilt parent assessment scale is designed to measure the severity of ADHD symptoms for children aged 6 to 12. It has 2 components: symptom assessment and impairment in performance. The symptom assessment screens for symptoms relevant to inattentive (items 1-9) and hyperactive (items 10-18) ADHD. The items 49-56 are performance measures. The symptom measures in the scale, scored 0 to 3. A positive response in symptom assessment part is a 2 or 3 (often, very often). The performance measures in the scale, scored 1 to 5, with 4 and 5 being somewhat of a problem/problematic.
  The scoring standard for ADHD Combined Inattention/Hyperactivity: Must score a 2 or 3 on 6 out of 9 items not only on questions 1-9 but also on questions 10-18. AND Score a 4 or 5 on any of the Performance questions 49-56. The higher scores mean a worse outcome.
The changes in ADHD clinical symptoms-ADHD Combined Inattention/Hyperactivity estimated by Chinese version of Vanderbilt teacher assessment scale | at baseline
  The Vanderbilt teacher assessment scale is designed to measure the severity of ADHD symptoms for children aged 6 to 12. It has 2 components: symptom assessment and impairment in performance. The symptom assessment screens for symptoms relevant to inattentive (items 1-9) and hyperactive (items 10-18) ADHD. The items 36-43 are performance measures. The symptom measures in the scale, scored 0 to 3. A positive response in symptom assessment part is a 2 or 3 (often, very often). The performance measures in the scale, scored 1 to 5, with 4 and 5 being somewhat of a problem/problematic.
  The scoring standard for ADHD Combined Inattention/Hyperactivity: Must score a 2 or 3 on 6 out of 9 items not only on questions 1-9 but also on questions 10-18. AND Score a 4 or 5 on any of the Performance questions 36-43. The higher scores mean a worse outcome.
The changes in ADHD clinical symptoms-Predominantly Inattentive subtype estimated by Chinese version of Vanderbilt parent follow-up assessment | at weeks 4 and 8
  The Vanderbilt parent follow-up assessment is designed to track treatment effect over time for ADHD children aged 6 to 12. It has 2 components: symptom assessment and impairment in performance. The symptom assessment screens for symptoms relevant to inattentive (items 1-9) and hyperactive (items 10-18) ADHD. The items 19-26 are performance measures. The symptom measures in the scale, scored 0 to 3 (Never, Occasionally, Often, Very Often). The performance measures in the scale, scored 1 to 5 (Excellent, Above Average, Average, Somewhat of a Problem, Performance Problematic).
  The scoring standard for Predominantly Inattentive subtype: 1) Calculate Total Symptom Score for questions 1-18. 2) Calculate Average Performance Score for questions 19-26. The higher scores mean a worse outcome.
The changes in ADHD clinical symptoms-Predominantly Inattentive subtype estimated by Chinese version of Vanderbilt teacher follow-up assessment | at weeks 4 and 8
  The Vanderbilt teacher follow-up assessment is designed to track treatment effect over time for ADHD children aged 6 to 12. It has 2 components: symptom assessment and impairment in performance. The symptom assessment screens for symptoms relevant to inattentive (items 1-9) and hyperactive (items 10-18) ADHD. The items 19-26 are performance measures. The symptom measures in the scale, scored 0 to 3 (Never, Occasionally, Often, Very Often). The performance measures in the scale, scored 1 to 5 (Excellent, Above Average, Average, Somewhat of a Problem, Performance Problematic).
  The scoring standard for Predominantly Inattentive subtype: 1) Calculate Total Symptom Score for questions 1-18. 2) Calculate Average Performance Score for questions 19-26. The higher scores mean a worse outcome.
The changes in ADHD clinical symptoms-Predominantly Hyperactive/Impulsive subtype estimated by Chinese version of Vanderbilt parent follow-up assessment | at weeks 4 and 8
  The Vanderbilt parent follow-up assessment is designed to track treatment effect over time for ADHD children aged 6 to 12. It has 2 components: symptom assessment and impairment in performance. The symptom assessment screens for symptoms relevant to inattentive (items 1-9) and hyperactive (items 10-18) ADHD. The items 19-26 are performance measures. The symptom measures in the scale, scored 0 to 3 (Never, Occasionally, Often, Very Often). The performance measures in the scale, scored 1 to 5 (Excellent, Above Average, Average, Somewhat of a Problem, Performance Problematic).
  The scoring standard for Predominantly Hyperactive/Impulsive subtype: 1) Calculate Total Symptom Score for questions 1-18. 2) Calculate Average Performance Score for questions 19-26. The higher scores mean a worse outcome.
The changes in ADHD clinical symptoms-Predominantly Hyperactive/Impulsive subtype estimated by Chinese version of Vanderbilt teacher follow-up assessment | at weeks 4 and 8
  The Vanderbilt teacher follow-up assessment is designed to track treatment effect over time for ADHD children aged 6 to 12. It has 2 components: symptom assessment and impairment in performance. The symptom assessment screens for symptoms relevant to inattentive (items 1-9) and hyperactive (items 10-18) ADHD. The items 19-26 are performance measures. The symptom measures in the scale, scored 0 to 3 (Never, Occasionally, Often, Very Often). The performance measures in the scale, scored 1 to 5 (Excellent, Above Average, Average, Somewhat of a Problem, Performance Problematic).
  The scoring standard for Predominantly Hyperactive/Impulsive subtype: 1) Calculate Total Symptom Score for questions 1-18. 2) Calculate Average Performance Score for questions 19-26. The higher scores mean a worse outcome.
The changes in ADHD clinical symptoms-ADHD Combined Inattention/Hyperactivity estimated by Chinese version of Vanderbilt parent follow-up assessment | at weeks 4 and 8
  The Vanderbilt parent follow-up assessment is designed to track treatment effect over time for ADHD children aged 6 to 12. It has 2 components: symptom assessment and impairment in performance. The symptom assessment screens for symptoms relevant to inattentive (items 1-9) and hyperactive (items 10-18) ADHD. The items 19-26 are performance measures. The symptom measures in the scale, scored 0 to 3 (Never, Occasionally, Often, Very Often). The performance measures in the scale, scored 1 to 5 (Excellent, Above Average, Average, Somewhat of a Problem, Performance Problematic).
  The scoring standard for ADHD Combined Inattention/Hyperactivity: 1) Calculate Total Symptom Score for questions 1-18. 2) Calculate Average Performance Score for questions 19-26. The higher scores mean a worse outcome.
The changes in ADHD clinical symptoms-ADHD Combined Inattention/Hyperactivity estimated by Chinese version of Vanderbilt teacher follow-up assessment | at weeks 4 and 8
  The Vanderbilt teacher follow-up assessment is designed to track treatment effect over time for ADHD children aged 6 to 12. It has 2 components: symptom assessment and impairment in performance. The symptom assessment screens for symptoms relevant to inattentive (items 1-9) and hyperactive (items 10-18) ADHD. The items 19-26 are performance measures. The symptom measures in the scale, scored 0 to 3 (Never, Occasionally, Often, Very Often). The performance measures in the scale, scored 1 to 5 (Excellent, Above Average, Average, Somewhat of a Problem, Performance Problematic).
  The scoring standard for ADHD Combined Inattention/Hyperactivity: 1) Calculate Total Symptom Score for questions 1-18. 2) Calculate Average Performance Score for questions 19-26. The higher scores mean a worse outcome.
The changes in ADHD clinical symptoms | at baseline, weeks 4 and 8
  The Questionnaire - Children with Difficulties (QCD) measures the daily-life problems in children aged 6-18 years during the special time of the day, including in the morning, during school, after school, in the evening, and overall difficulties over the entire day and night. It has been proved the Chinese version of QCD has good validity and reliability. Filled in by the parents, the scale consists of 20 questions with regard to ADHD-related difficulties. Each question is scored on a four-point scale: 0 = completely disagree, 1 = somewhat (partially) agree, 2 = mostly agree, and 3 = completely agree. Score of 30 - 35 is considered as cut-off value for functional impairment and score of less than 30 is considered as functional impairment (Full marks: 57). The lower scores indicate lower life functioning and more difficulty in children's daily activities.

SECONDARY OUTCOMES:
Serum concentration of vitamin A. | at baseline and weeks 8
  Vitamin A state is measured by the serum concentration of retinol through high performance liquid chromatography (HPLC) from 2 milliliter of venous blood. The vitamin A status is categorized based on serum retinol: <0.35 µmol/L is considered very deficient, 0.35-0.7 µmol/L deficient, 0.7-1.05 µmol/L marginal, 1.05-2.56 µmol/L adequate, and >2.56 µmol/L toxic. Too low or too high concentrations are harmful
Serum concentration of vitamin D. | at baseline and weeks 8
  Vitamin D state is measured by the serum concentration of 25OHD through high performance liquid chromatography (HPLC) from 2 milliliter of venous blood. The values of serum vitamin D level are classified into 4 categories: <30 nmol/L is regarded as deficiency, 30-50 nmol/L insufficiency, 50-250 nmol/L normal, and >250 nmol/L toxic . Too low or too high concentrations are harmful。

CONTACTS AND LOCATIONS:
Overall Officials: Li Chen, doctor, Study Director — Children's Hospital of Chongqing Medical University; yu T Li, MS, Study Chair — Children's Hospital of Chongqing Medical University
Locations (3):
- China (3):
  - Growth, Development and Mental health of Children and Adolescence Center, Chongqing, Chongqing Municipality
  - the First Hospital of Jilin University, Changchun, Jilin
  - Qilu Hospital of Shandong University, Jinan, Shandonng

IPD SHARING:
Plan to Share IPD: No
Data is confidential during the study.

REFERENCES:
- [Background] Dehbokri N, Noorazar G, Ghaffari A, Mehdizadeh G, Sarbakhsh P, Ghaffary S. Effect of vitamin D treatment in children with attention-deficit hyperactivity disorder. World J Pediatr. 2019 Feb;15(1):78-84. doi: 10.1007/s12519-018-0209-8. Epub 2018 Nov 19. PMID 30456564
- [Background] Elshorbagy HH, Barseem NF, Abdelghani WE, Suliman HAI, Al-Shokary AH, Abdulsamea SE, Elsadek AE, Abdel Maksoud YH, Nour El Din DMAE. Impact of Vitamin D Supplementation on Attention-Deficit Hyperactivity Disorder in Children. Ann Pharmacother. 2018 Jul;52(7):623-631. doi: 10.1177/1060028018759471. Epub 2018 Feb 18. PMID 29457493
- [Background] Evans E, Piccio L, Cross AH. Use of Vitamins and Dietary Supplements by Patients With Multiple Sclerosis: A Review. JAMA Neurol. 2018 Aug 1;75(8):1013-1021. doi: 10.1001/jamaneurol.2018.0611. PMID 29710293
- [Background] Faraone SV. The pharmacology of amphetamine and methylphenidate: Relevance to the neurobiology of attention-deficit/hyperactivity disorder and other psychiatric comorbidities. Neurosci Biobehav Rev. 2018 Apr;87:255-270. doi: 10.1016/j.neubiorev.2018.02.001. Epub 2018 Feb 8. PMID 29428394
- [Background] Fasihpour B, Moayeri H, Shariat M, Keihanidoust Z, Effatpanah M, Khedmat L. Vitamin D deficiency in school-age Iranian children with attention-deficit/hyperactivity disorder (ADHD) symptoms: A critical comparison with healthy controls. Child Neuropsychol. 2020 May;26(4):460-474. doi: 10.1080/09297049.2019.1665638. Epub 2019 Sep 13. PMID 31514566
- [Background] Fragoso YD, Stoney PN, McCaffery PJ. The evidence for a beneficial role of vitamin A in multiple sclerosis. CNS Drugs. 2014 Apr;28(4):291-9. doi: 10.1007/s40263-014-0148-4. PMID 24557746
- [Background] Gallo EF, Posner J. Moving towards causality in attention-deficit hyperactivity disorder: overview of neural and genetic mechanisms. Lancet Psychiatry. 2016 Jun;3(6):555-67. doi: 10.1016/S2215-0366(16)00096-1. Epub 2016 May 13. PMID 27183902
- [Background] Hinshaw SP. Attention Deficit Hyperactivity Disorder (ADHD): Controversy, Developmental Mechanisms, and Multiple Levels of Analysis. Annu Rev Clin Psychol. 2018 May 7;14:291-316. doi: 10.1146/annurev-clinpsy-050817-084917. Epub 2017 Dec 8. PMID 29220204
- [Background] Lopes FM, da Motta LL, De Bastiani MA, Pfaffenseller B, Aguiar BW, de Souza LF, Zanatta G, Vargas DM, Schonhofen P, Londero GF, de Medeiros LM, Freire VN, Dafre AL, Castro MA, Parsons RB, Klamt F. RA Differentiation Enhances Dopaminergic Features, Changes Redox Parameters, and Increases Dopamine Transporter Dependency in 6-Hydroxydopamine-Induced Neurotoxicity in SH-SY5Y Cells. Neurotox Res. 2017 May;31(4):545-559. doi: 10.1007/s12640-016-9699-0. Epub 2017 Feb 2. PMID 28155214
- [Background] McCaffery P, Drager UC. High levels of a retinoic acid-generating dehydrogenase in the meso-telencephalic dopamine system. Proc Natl Acad Sci U S A. 1994 Aug 2;91(16):7772-6. doi: 10.1073/pnas.91.16.7772. PMID 8052659
- [Background] Mohammadpour N, Jazayeri S, Tehrani-Doost M, Djalali M, Hosseini M, Effatpanah M, Davari-Ashtiani R, Karami E. Effect of vitamin D supplementation as adjunctive therapy to methylphenidate on ADHD symptoms: A randomized, double blind, placebo-controlled trial. Nutr Neurosci. 2018 Apr;21(3):202-209. doi: 10.1080/1028415X.2016.1262097. Epub 2016 Dec 7. PMID 27924679
- [Background] Moretti R, Morelli ME, Caruso P. Vitamin D in Neurological Diseases: A Rationale for a Pathogenic Impact. Int J Mol Sci. 2018 Jul 31;19(8):2245. doi: 10.3390/ijms19082245. PMID 30065237
- [Background] Ono K, Yamada M. Vitamin A and Alzheimer's disease. Geriatr Gerontol Int. 2012 Apr;12(2):180-8. doi: 10.1111/j.1447-0594.2011.00786.x. Epub 2011 Dec 23. PMID 22221326
- [Background] Palacios C, Gonzalez L. Is vitamin D deficiency a major global public health problem? J Steroid Biochem Mol Biol. 2014 Oct;144 Pt A:138-45. doi: 10.1016/j.jsbmb.2013.11.003. Epub 2013 Nov 12. PMID 24239505
- [Background] Pertile RA, Cui X, Eyles DW. Vitamin D signaling and the differentiation of developing dopamine systems. Neuroscience. 2016 Oct 1;333:193-203. doi: 10.1016/j.neuroscience.2016.07.020. Epub 2016 Jul 20. PMID 27450565
- [Background] Pertile RAN, Cui X, Hammond L, Eyles DW. Vitamin D regulation of GDNF/Ret signaling in dopaminergic neurons. FASEB J. 2018 Feb;32(2):819-828. doi: 10.1096/fj.201700713R. Epub 2018 Jan 4. PMID 29018141
- [Background] Russell VA. Overview of animal models of attention deficit hyperactivity disorder (ADHD). Curr Protoc Neurosci. 2011 Jan;Chapter 9:Unit9.35. doi: 10.1002/0471142301.ns0935s54. PMID 21207367
- [Background] Seyedi M, Gholami F, Samadi M, Djalali M, Effatpanah M, Yekaninejad MS, Hashemi R, Abdolahi M, Chamari M, Honarvar NM. The Effect of Vitamin D3 Supplementation on Serum BDNF, Dopamine, and Serotonin in Children with Attention-Deficit/Hyperactivity Disorder. CNS Neurol Disord Drug Targets. 2019;18(6):496-501. doi: 10.2174/1871527318666190703103709. PMID 31269890
- [Background] Song P, Wang J, Wei W, Chang X, Wang M, An L. The Prevalence of Vitamin A Deficiency in Chinese Children: A Systematic Review and Bayesian Meta-Analysis. Nutrients. 2017 Nov 25;9(12):1285. doi: 10.3390/nu9121285. PMID 29186832
- [Background] Duric NS, Assmus J, Gundersen D, Duric Golos A, Elgen IB. Multimodal treatment in children and adolescents with attention-deficit/hyperactivity disorder: a 6-month follow-up. Nord J Psychiatry. 2017 Jul;71(5):386-394. doi: 10.1080/08039488.2017.1305446. Epub 2017 Mar 27. PMID 28345387
- [Background] Biederman J, Faraone SV. Attention-deficit hyperactivity disorder. Lancet. 2005 Jul 16-22;366(9481):237-48. doi: 10.1016/S0140-6736(05)66915-2. PMID 16023516
- [Background] Wolraich ML, Hagan JF Jr, Allan C, Chan E, Davison D, Earls M, Evans SW, Flinn SK, Froehlich T, Frost J, Holbrook JR, Lehmann CU, Lessin HR, Okechukwu K, Pierce KL, Winner JD, Zurhellen W; SUBCOMMITTEE ON CHILDREN AND ADOLESCENTS WITH ATTENTION-DEFICIT/HYPERACTIVE DISORDER. Clinical Practice Guideline for the Diagnosis, Evaluation, and Treatment of Attention-Deficit/Hyperactivity Disorder in Children and Adolescents. Pediatrics. 2019 Oct;144(4):e20192528. doi: 10.1542/peds.2019-2528. PMID 31570648
- [Derived] Zhou P, Wolraich ML, Cao AH, Jia FY, Liu B, Zhu L, Liu Y, Li X, Li C, Peng B, Yang T, Chen J, Cheng Q, Li T, Chen L. Adjuvant effects of vitamin A and vitamin D supplementation on treatment of children with attention-deficit/hyperactivity disorder: a study protocol for a randomised, double-blinded, placebo-controlled, multicentric trial in China. BMJ Open. 2021 Jun 16;11(6):e050541. doi: 10.1136/bmjopen-2021-050541. PMID 34135055